CLINICAL TRIAL: NCT00998985
Title: A Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Grazoprevir (MK-5172) in Hepatitis C Infected Male Patients
Brief Title: A Study of Grazoprevir (MK-5172) in Hepatitis C-Infected Male Participants (MK-5172-004)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5172-004; 2009_678 (Other: Merck); 2009-015563-13 (EudraCT Number)
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Results first posted 2016-03-02 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-06

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — grazoprevir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (14):
- 400 mg Grazoprevir - GT1 (Experimental): GT1 HCV-infected Participants: 400 mg Grazoprevir or Placebo
  Interventions: Drug: Grazoprevir; Drug: Placebo
- 600 mg Grazoprevir - GT1 (Experimental): GT1 HCV-infected Participants: 600 mg Grazoprevir or Placebo
  Interventions: Drug: Grazoprevir; Drug: Placebo
- 800 mg Grazoprevir - GT1 (Experimental): GT1 HCV-infected Participants: 800 mg Grazoprevir or Placebo
  Interventions: Drug: Grazoprevir; Drug: Placebo
- 400 mg Grazoprevir - GT3 (Experimental): GT3 HCV-infected Participants: 400 mg Grazoprevir or Placebo
  Interventions: Drug: Grazoprevir; Drug: Placebo
- 600 mg Grazoprevir - GT3 (Experimental): GT3 HCV-infected Participants: 600 mg Grazoprevir or Placebo
  Interventions: Drug: Grazoprevir; Drug: Placebo
- 800 mg Grazoprevir - GT3 (Experimental): GT3 HCV-infected Participants: 800 mg Grazoprevir or Placebo
  Interventions: Drug: Grazoprevir; Drug: Placebo
- 200 mg Grazoprevir - GT1 (Experimental): GT1 HCV-infected Participants: 200 mg Grazoprevir or Placebo
  Interventions: Drug: Grazoprevir; Drug: Placebo
- 100 mg Grazoprevir - GT1 (Experimental): GT1 HCV-infected Participants: 100 mg Grazoprevir or Placebo
  Interventions: Drug: Grazoprevir; Drug: Placebo
- 50 mg Grazoprevir - GT1 (Experimental): GT1 HCV-infected Participants: 50 mg Grazoprevir or Placebo
  Interventions: Drug: Grazoprevir; Drug: Placebo
- 200 mg Grazoprevir - GT3 (Experimental): GT3 HCV-infected Participants: 200 mg Grazoprevir or Placebo
  Interventions: Drug: Grazoprevir; Drug: Placebo
- 100 mg Grazoprevir - GT3 (Experimental): GT3 HCV-infected Participants: 100 mg Grazoprevir or Placebo
  Interventions: Drug: Grazoprevir; Drug: Placebo
- 50 mg Grazoprevir - GT3 (Experimental): GT3 HCV-infected Participants: 50 mg Grazoprevir or Placebo
  Interventions: Drug: Grazoprevir; Drug: Placebo
- 30 mg Grazoprevir - GT1 (Experimental): GT1 HCV-infected Participants: 30 mg Grazoprevir or Placebo
  Interventions: Drug: Grazoprevir; Drug: Placebo
- 10 mg Grazoprevir - GT1 (Experimental): GT1 HCV-infected Participants: 10 mg Grazoprevir or Placebo
  Interventions: Drug: Grazoprevir; Drug: Placebo

INTERVENTIONS:
Drug: Grazoprevir — 10, 30, 50, 100, 200, 400, 600 or 800 mg Grazoprevir tablets, orally, once a day for 7 days
Drug: Placebo — Placebo tablet, orally, once a day for 7 days

SUMMARY:
This multiple dose study will assess the safety, tolerability, pharmacokinetics and pharmacodynamics of grazoprevir (MK-5172) in Genotype (GT) 1 and GT3 Hepatitis C virus (HCV)- infected participants. The primary hypothesis is that administration of grazoprevir for 7 days is sufficiently safe and well tolerated in HCV-infected males.

ELIGIBILITY:
Inclusion Criteria:

* Baseline health is stable.
* Has a clinical diagnosis of chronic HCV infection.

Exclusion Criteria:

* Has a history of stroke or chronic seizures.
* Has a history of cancer.
* Has a history of human immunodeficiency virus (HIV) infection.
* Has had major surgery, donated blood or participated in another investigational study within the past 3 months.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2010-02-23 (Actual); Primary Completion 2012-11-08 (Actual); Study Completion 2012-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Yeh WW, Fraser IP, Jumes P, Petry A, Lepeleire I, Robberechts M, Reitmann C, Van Dyck K, Huang X, Guo Z, Panebianco D, Nachbar RB, O'Mara E, Wagner JA, Butterton JR, Dutko FJ, Moiseev V, Kobalava Z, Huser A, Visan S, Schwabe C, Gane E, Popa S, Ghicavii N, Uhle M, Wagner F. Antiviral Activity, Safety, and Tolerability of Multiple Ascending Doses of Elbasvir or Grazoprevir in Participants Infected With Hepatitis C Virus Genotype-1 or -3. Clin Ther. 2018 May;40(5):704-718.e6. doi: 10.1016/j.clinthera.2018.03.002. Epub 2018 Apr 25. PMID 29703432
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=5172-004&kw=5172-004&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One of the originally planned treatment groups (50 mg Grazoprevir - GT3) was not conducted because other results indicated that further evaluation of 50 mg Grazoprevir in GT3 participants was not necessary. It is therefore not included in the Participant Flow.
Groups:
- 400 mg Grazoprevir - GT1: GT1 HCV-infected Participants: 400 mg Grazoprevir orally, once daily for 7 consecutive days
- 600 mg Grazoprevir - GT1: GT1 HCV-infected Participants: 600 mg Grazoprevir orally, once daily for 7 consecutive days
- 800 mg Grazoprevir - GT1: GT1 HCV-infected Participants: 800 mg Grazoprevir orally, once daily for 7 consecutive days
- 400 mg Grazoprevir - GT3: GT3 HCV-infected Participants: 400 mg Grazoprevir orally, once daily for 7 consecutive days
- 600 mg Grazoprevir - GT3: GT3 HCV-infected Participants: 600 mg Grazoprevir orally, once daily for 7 consecutive days
- 800 mg Grazoprevir - GT3: GT3 HCV-infected Participants: 800 mg Grazoprevir orally, once daily for 7 consecutive days
- 200 mg Grazoprevir - GT1: GT1 HCV-infected Participants: 200 mg Grazoprevir orally, once daily for 7 consecutive days
- 100 mg Grazoprevir - GT1: GT1 HCV-infected Participants: 100 mg Grazoprevir orally, once daily for 7 consecutive days
- 50 mg Grazoprevir - GT1: GT1 HCV-infected Participants: 50 mg Grazoprevir orally, once daily for 7 consecutive days
- 200 mg Grazoprevir - GT3: GT3 HCV-infected Participants: 200 mg Grazoprevir orally, once daily for 7 consecutive days
- 100 mg Grazoprevir - GT3: GT3 HCV-infected Participants: 100 mg Grazoprevir orally, once daily for 7 consecutive days
- 30 mg Grazoprevir - GT1: GT1 HCV-infected Participants: 30 mg Grazoprevir orally, once daily for 7 consecutive days
- 10 mg Grazoprevir - GT1: GT1 HCV-infected Participants: 10 mg Grazoprevir orally, once daily for 7 consecutive days
- Placebo for Grazoprevir - GT1 and GT3: GT1 and GT3 HCV-infected Participants: Placebo for Grazoprevir orally, once daily for 7 consecutive days
Period: Overall Study
Arm/Group | 400 mg Grazoprevir - GT1 | 600 mg Grazoprevir - GT1 | 800 mg Grazoprevir - GT1 | 400 mg Grazoprevir - GT3 | 600 mg Grazoprevir - GT3 | 800 mg Grazoprevir - GT3 | 200 mg Grazoprevir - GT1 | 100 mg Grazoprevir - GT1 | 50 mg Grazoprevir - GT1 | 200 mg Grazoprevir - GT3 | 100 mg Grazoprevir - GT3 | 30 mg Grazoprevir - GT1 | 10 mg Grazoprevir - GT1 | Placebo for Grazoprevir - GT1 and GT3
Started | 5 | 5 | 15 | 5 | 5 | 5 | 5 | 5 | 6 | 5 | 5 | 5 | 5 | 15
Completed | 5 | 5 | 15 | 5 | 5 | 4 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 15
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | 400 mg Grazoprevir - GT1 | 600 mg Grazoprevir - GT1 | 800 mg Grazoprevir - GT1 | 400 mg Grazoprevir - GT3 | 600 mg Grazoprevir - GT3 | 800 mg Grazoprevir - GT3 | 200 mg Grazoprevir - GT1 | 100 mg Grazoprevir - GT1 | 50 mg Grazoprevir - GT1 | 200 mg Grazoprevir - GT3 | 100 mg Grazoprevir - GT3 | 30 mg Grazoprevir - GT1 | 10 mg Grazoprevir - GT1 | Placebo for Grazoprevir - GT1 and GT3 | Total
Number analyzed (Participants) | 5 | 5 | 15 | 5 | 5 | 5 | 5 | 5 | 6 | 5 | 5 | 5 | 5 | 15 | 91
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.4 (12.8) | 47.2 (12.2) | 46.7 (9.7) | 42.8 (14.4) | 38.0 (13.1) | 46.2 (10.8) | 51.0 (16.2) | 48.4 (5.9) | 36.8 (6.0) | 40.0 (10.2) | 31.4 (6.3) | 55.8 (5.4) | 48.4 (13.1) | 45.6 (11.5) | 44.7 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 5 | 5 | 15 | 5 | 5 | 5 | 5 | 5 | 6 | 5 | 5 | 5 | 5 | 15 | 91

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical and Laboratory Adverse Events (AEs)
Description: An AE is any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR's product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the SPONSOR's product, is also an AE.
Time Frame: All AEs: 15 Days after last dose; Serious AEs (SAEs) up to 2 months after last dose (Up to 67 days)
Population: All participants who received at least one dose of the investigational drug according to the treatment(s) they actually received. Participants with either GT1 or GT3 who received the same treatment were combined for the summary into a single GT1 and GT3 arm.
Measure: Number; unit: Participants
Groups:
- 400 mg Grazoprevir - GT1 and GT3: GT1 and GT3 HCV-infected Participants: 400 mg Grazoprevir orally, once daily for 7 consecutive days
- 600 mg Grazoprevir - GT1 and GT3: GT1 and GT3 HCV-infected Participants: 600 mg Grazoprevir orally, once daily for 7 consecutive days
- 800 mg Grazoprevir - GT1 and GT3: GT1 and GT3 HCV-infected Participants: 800 mg Grazoprevir orally, once daily for 7 consecutive days
- 200 mg Grazoprevir - GT1 and GT3: GT1 and GT3 HCV-infected Participants: 200 mg Grazoprevir orally, once daily for 7 consecutive days
- 100 mg Grazoprevir - GT1 and GT3: GT1 and GT3 HCV-infected Participants: 100 mg Grazoprevir orally, once daily for 7 consecutive days
Arm/Group | 400 mg Grazoprevir - GT1 and GT3 | 600 mg Grazoprevir - GT1 and GT3 | 800 mg Grazoprevir - GT1 and GT3 | 200 mg Grazoprevir - GT1 and GT3 | 100 mg Grazoprevir - GT1 and GT3 | 50 mg Grazoprevir - GT1 | 30 mg Grazoprevir - GT1 | 10 mg Grazoprevir - GT1 | Placebo for Grazoprevir - GT1 and GT3
Number analyzed (Participants) | 10 | 10 | 20 | 10 | 10 | 6 | 5 | 5 | 15
Participants | 6 | 3 | 13 | 4 | 1 | 0 | 3 | 4 | 2

2. Secondary Outcome: Area Under the Curve for 0 to 24 Hours Post-dose (AUC[0-24hr]) of Grazoprevir on Day 7
Description: Blood samples were collected on Day 7 at pre-dose up to 24 hours post-dose in order to determine the AUC 0-24hrs of Grazoprevir. It is hypothesized that the Geometric Mean of Day 7 Grazoprevir AUC0-24hr. exceeds 3.2 uM.hr.
Time Frame: Day 7 at the following time points: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, and 24 hours post-dose
Population: Participants who complied with the protocol sufficiently to ensure that these data will exhibit the effects of treatment, according to the underlying scientific model. GT1 or GT3 participants who received the same treatment were combined into a single arm. Participants with placebo were not analyzed as they did not receive grazoprevir.
Measure: Geometric Mean (90% Confidence Interval); unit: uM.hr
Arm/Group | 400 mg Grazoprevir - GT1 and GT3 | 600 mg Grazoprevir - GT1 and GT3 | 800 mg Grazoprevir - GT1 and GT3 | 200 mg Grazoprevir - GT1 and GT3 | 100 mg Grazoprevir - GT1 and GT3 | 50 mg Grazoprevir - GT1 | 30 mg Grazoprevir - GT1 | 10 mg Grazoprevir - GT1 | Placebo for Grazoprevir - GT1 and GT3
Number analyzed (Participants) | 10 | 10 | 18 | 10 | 10 | 5 | 5 | 5 | 0
uM.hr | 18.2 [12.2 to 27.2] | 41.9 [28.0 to 62.6] | 72.5 [54.1 to 97.2] | 3.21 [2.14 to 4.80] | 1.16 [0.774 to 1.73] | 0.419 [0.237 to 0.740] | 0.260 [0.147 to 0.459] | 0.0628 [0.0355 to 0.111] |

3. Secondary Outcome: 24 Hour Plasma Concentration (C[24hr]) of Grazoprevir on Day 7
Description: Blood samples were collected on Day 7 at 24 hours post-dose in order to determine the C24hr of Grazoprevir. It is hypothesized that the Geometric Mean of Day 7 Grazoprevir C24hr exceeds 28 nM.
Time Frame: Day 7 at 24 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (90% Confidence Interval); unit: nM
Arm/Group | 400 mg Grazoprevir - GT1 and GT3 | 600 mg Grazoprevir - GT1 and GT3 | 800 mg Grazoprevir - GT1 and GT3 | 200 mg Grazoprevir - GT1 and GT3 | 100 mg Grazoprevir - GT1 and GT3 | 50 mg Grazoprevir - GT1 | 30 mg Grazoprevir - GT1 | 10 mg Grazoprevir - GT1 | Placebo for Grazoprevir - GT1 and GT3
Number analyzed (Participants) | 10 | 10 | 18 | 10 | 10 | 5 | 5 | 5 | 0
nM | 70.2 [46.9 to 105] | 93.2 [62.3 to 140] | 174 [130 to 233] | 22.2 [14.8 to 33.2] | 20.1 [13.4 to 30.1] | 12.7 [7.16 to 22.4] | 7.20 [4.07 to 12.7] | 2.41 [1.36 to 4.27] |

4. Secondary Outcome: Maximum log10 HCV RNA Reduction From Baseline Following Administration of Grazoprevir in Participants With GT1 HCV or Pooled GT1 and GT3 HCV Participants Treated With Placebo
Description: Blood samples were collected at baseline and at intervals up to 2 months post-dose in order to determine the maximum log10 reduction from baseline in plasma HCV RNA, expressed in international units (IU)/mL.
Time Frame: Baseline and up to approximately 2 months
Population: Participants who complied with the protocol sufficiently to ensure that these data will exhibit the effects of treatment, according to the underlying scientific model. One GT1 participant treated with 50 mg grazoprevir, who discontinued, and all GT3 participants treated with grazoprevir were excluded from analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 IU/mL
Groups:
- Placebo for Grazoprevir - GT1 and GT3: Pooled GT1 and GT3 HCV-infected Participants: Placebo for Grazoprevir orally, once daily for 7 consecutive days
Arm/Group | 400 mg Grazoprevir - GT1 | 600 mg Grazoprevir - GT1 | 800 mg Grazoprevir - GT1 | 200 mg Grazoprevir - GT1 | 100 mg Grazoprevir - GT1 | 50 mg Grazoprevir - GT1 | 30 mg Grazoprevir - GT1 | 10 mg Grazoprevir - GT1 | Placebo for Grazoprevir - GT1 and GT3 | 400 mg Grazoprevir - GT3 | 600 mg Grazoprevir - GT3 | 800 mg Grazoprevir - GT3 | 200 mg Grazoprevir - GT3 | 100 mg Grazoprevir - GT3
Number analyzed (Participants) | 5 | 5 | 15 | 5 | 5 | 5 | 5 | 5 | 15 | 0 | 0 | 0 | 0 | 0
log10 IU/mL | 5.14 [4.55 to 5.73] | 5.32 [4.73 to 5.91] | 5.72 [5.38 to 6.07] | 5.53 [4.94 to 6.12] | 4.74 [4.15 to 5.33] | 5.26 [4.67 to 5.85] | 5.06 [4.47 to 5.66] | 3.84 [3.25 to 4.43] | 0.39 [0.04 to 0.73] |  |  |  |  |
Statistical Analysis 1: Comparison: 10 mg Grazoprevir - GT1 vs Placebo for Grazoprevir - GT1 and GT3; It is hypothesized that one or more doses of Grazoprevir will reduce GT1 viral load by at least 3 log10; Test type: Superiority or Other; Least Squares Mean (LSM) Difference = 3.46, 90% CI 2-sided [2.89 to 4.03] — LSM Difference (grazoprevir-placebo) and confidence intervals from ANOVA model with maximum log10 HCV reduction as response and a fixed effect for treatment
Statistical Analysis 2: Comparison: 30 mg Grazoprevir - GT1 vs Placebo for Grazoprevir - GT1 and GT3; It is hypothesized that one or more doses of Grazoprevir will reduce GT1 viral load by at least 3 log10; Test type: Superiority or Other; LSM Difference = 4.68, 90% CI 2-sided [4.11 to 5.25] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: 50 mg Grazoprevir - GT1 vs Placebo for Grazoprevir - GT1 and GT3; It is hypothesized that one or more doses of Grazoprevir will reduce GT1 viral load by at least 3 log10; Test type: Superiority or Other; LSM Difference = 4.87, 90% CI 2-sided [4.30 to 5.44] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: 100 mg Grazoprevir - GT1 vs Placebo for Grazoprevir - GT1 and GT3; It is hypothesized that one or more doses of Grazoprevir will reduce GT1 viral load by at least 3 log10; Test type: Superiority or Other; LSM Difference = 4.35, 90% CI 2-sided [3.78 to 4.92] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: 200 mg Grazoprevir - GT1 vs Placebo for Grazoprevir - GT1 and GT3; It is hypothesized that one or more doses of Grazoprevir will reduce GT1 viral load by at least 3 log10; Test type: Superiority or Other; LSM Difference = 5.15, 90% CI 2-sided [4.58 to 5.72] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: 400 mg Grazoprevir - GT1 vs Placebo for Grazoprevir - GT1 and GT3; It is hypothesized that one or more doses of Grazoprevir will reduce GT1 viral load by at least 3 log10; Test type: Superiority or Other; LSM Difference = 4.76, 90% CI 2-sided [4.19 to 5.33] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 7: Comparison: 600 mg Grazoprevir - GT1 vs Placebo for Grazoprevir - GT1 and GT3; It is hypothesized that one or more doses of Grazoprevir will reduce GT1 viral load by at least 3 log10; Test type: Superiority or Other; LSM Difference = 4.93, 90% CI 2-sided [4.36 to 5.50] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 8: Comparison: 800 mg Grazoprevir - GT1 vs Placebo for Grazoprevir - GT1 and GT3; It is hypothesized that one or more doses of Grazoprevir will reduce GT1 viral load by at least 3 log10; Test type: Superiority or Other; LSM Difference = 5.34, 90% CI 2-sided [4.93 to 5.74] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Maximum log10 HCV RNA Reduction From Baseline Following Administration of Grazoprevir in Participants With GT3 HCV or Pooled GT1 and GT3 HCV Participants Treated With Placebo
Description: Blood samples were collected at baseline and at intervals up to 2 months post-dose in order to determine the maximum log10 reduction from baseline in plasma HCV RNA.
Time Frame: Baseline and up to approximately 2 months
Population: Participants who complied with the protocol sufficiently to ensure that these data will exhibit the effects of treatment, according to the underlying scientific model. One GT3 participant treated with 800 mg grazoprevir, who discontinued, and all GT1 participants were excluded from analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 IU/mL
Arm/Group | 400 mg Grazoprevir - GT3 | 600 mg Grazoprevir - GT3 | 800 mg Grazoprevir - GT3 | 200 mg Grazoprevir - GT3 | 100 mg Grazoprevir - GT3 | Placebo for Grazoprevir - GT1 and GT3 | 800 mg Grazoprevir - GT1 | 600 mg Grazoprevir - GT1 | 400 mg Grazoprevir - GT1 | 200 mg Grazoprevir - GT1 | 100 mg Grazoprevir - GT1 | 50 mg Grazoprevir - GT1 | 30 mg Grazoprevir - GT1 | 10 mg Grazoprevir - GT1
Number analyzed (Participants) | 5 | 5 | 4 | 5 | 5 | 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
log10 IU/mL | 4.23 [3.65 to 4.81] | 5.36 [4.79 to 5.94] | 4.60 [3.95 to 5.24] | 3.32 [2.75 to 3.90] | 2.64 [2.06 to 3.22] | 0.39 [0.05 to 0.72] |  |  |  |  |  |  |  |
Statistical Analysis 1: Comparison: 100 mg Grazoprevir - GT3 vs Placebo for Grazoprevir - GT1 and GT3; It is hypothesized that one or more doses of Grazoprevir will reduce GT3 viral load by at least 2 log10; Test type: Superiority or Other; LSM Difference = 2.25, 90% CI 2-sided [1.70 to 2.81] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: 200 mg Grazoprevir - GT3 vs Placebo for Grazoprevir - GT1 and GT3; It is hypothesized that one or more doses of Grazoprevir will reduce GT3 viral load by at least 2 log10; Test type: Superiority or Other; LSM Difference = 2.94, 90% CI 2-sided [2.38 to 3.49] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: 400 mg Grazoprevir - GT3 vs Placebo for Grazoprevir - GT1 and GT3; It is hypothesized that one or more doses of Grazoprevir will reduce GT3 viral load by at least 2 log10; Test type: Superiority or Other; LSM Difference = 3.84, 90% CI 2-sided [3.29 to 4.40] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: 600 mg Grazoprevir - GT3 vs Placebo for Grazoprevir - GT1 and GT3; It is hypothesized that one or more doses of Grazoprevir will reduce GT3 viral load by at least 2 log10; Test type: Superiority or Other; LSM difference = 4.98, 90% CI 2-sided [4.42 to 5.53] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: 800 mg Grazoprevir - GT3 vs Placebo for Grazoprevir - GT1 and GT3; It is hypothesized that one or more doses of Grazoprevir will reduce GT3 viral load by at least 2 log10; Test type: Superiority or Other; LSM difference = 4.21, 90% CI 2-sided [3.60 to 4.81] — [estimate comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: All AEs: 15 Days after last dose; Serious AEs (SAEs) up to 2 months after last dose (Up to 67 days)
Description: All participants who received at least one dose of drug according to the treatment(s) they actually received. Participants with either GT1 or GT3 who received the same treatment are combined into a single GT1 and GT3 arm.
Arm/Group | 400 mg Grazoprevir - GT1 and GT3 | 600 mg Grazoprevir - GT1 and GT3 | 800 mg Grazoprevir - GT1 and GT3 | 200 mg Grazoprevir - GT1 and GT3 | 100 mg Grazoprevir - GT1 and GT3 | 50 mg Grazoprevir - GT1 | 30 mg Grazoprevir - GT1 | 10 mg Grazoprevir - GT1 | Placebo for Grazoprevir - GT1 and GT3
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/20 | 0/10 | 0/10 | 0/6 | 0/5 | 0/5 | 0/15
Other Adverse Events (participants affected / at risk) | 6/10 | 3/10 | 13/20 | 4/10 | 1/10 | 0/6 | 3/5 | 4/5 | 2/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 400 mg Grazoprevir - GT1 and GT3 (N=10) | 600 mg Grazoprevir - GT1 and GT3 (N=10) | 800 mg Grazoprevir - GT1 and GT3 (N=20) | 200 mg Grazoprevir - GT1 and GT3 (N=10) | 100 mg Grazoprevir - GT1 and GT3 (N=10) | 50 mg Grazoprevir - GT1 (N=6) | 30 mg Grazoprevir - GT1 (N=5) | 10 mg Grazoprevir - GT1 (N=5) | Placebo for Grazoprevir - GT1 and GT3 (N=15)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 6 (10) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (5) | 0 (0) | 8 (11) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (2)
Migraine (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.